CLINICAL TRIAL: NCT04991675
Title: The Role of Diaphragmatic Breathing Exercise on Urinary Incontinence Treatment: A Pilot Study
Brief Title: Diaphragmatic Breathing Exercises on Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: selva sen (Other)
Responsible Party: Sponsor-Investigator, selva sen, Research Assistant, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 126
Record Dates: First submitted 2021-07-02; First posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Urinary Incontinence
Keywords: Diaphragmatic breathing exercise; Pelvic floor muscles exercises; Kegel exercise; Urinary incontinence; Physiotherapy
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: Participants were randomized into two groups: pelvic floor muscle exercises (Group PFM n=20) and diaphragmatic breathing exercises (Group DB n=20). Exercise programs consisted of 1 set of contractions per day and each set included 30 repetitions for 6 weeks. Women were asked to complete forms of Incontinence Impact Questionnaire (IIQ-7) and the Urogenital Distress Inventory (UDI-6), Incontinence Quality of Life (I-QOL), and Overactive Bladder (OAB-V3) before starting the program and again at the end of the 6-week program. Changes from baseline were compared in both groups and between the two groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pelvic floor muscle exercises (Active Comparator): Exercises were taught in the supine position, as described by Kegel (1948), and it was confirmed that the women learned to use the correct muscles with vaginal palpation. During the exercise, the participants were informed not to pull the abdomen inwards, not to tighten their legs and hip muscles, and not move their pelvis.
  Interventions: Behavioral: pelvic floor muscle exercises
- diaphragmatic breathing exercises (Active Comparator): Diaphragmatic breathing exercise was taught in supine position. The movement of the symphysis pubis was examined to confirm that the pelvic floors' movement was also involved breathing. Abdominal palpation was used to elicit unawareness of the diaphragmatic breathing and to assess whether contractions were performed correctly.
  Interventions: Behavioral: diaphragmatic breathing exercises

INTERVENTIONS:
Behavioral: pelvic floor muscle exercises — During the first visit, the anatomy of the pelvic floor and the purpose of the program were explained. Exercises were taught in the supine position, as described by Kegel (1948), it was confirmed that the women learned to use the correct muscles with vaginal palpation. During the exercise, the participants were informed not to pull the abdomen inwards, not to tighten their legs and hip muscles, and not move their pelvis.
  Arms: pelvic floor muscle exercises
Behavioral: diaphragmatic breathing exercises — During the first visit, the anatomy of the diaphragm and abdominal wall and the purpose of the program were explained. Diaphragmatic breathing exercise was taught in supine position. The movement of the symphysis pubis was examined to confirm that the pelvic floors' movement was also involved breathing. Abdominal palpation was used to elicit unawareness of the diaphragmatic breathing and to assess whether contractions were performed correctly.
  Arms: diaphragmatic breathing exercises

SUMMARY:
The main aim of this pilot study was to examine the effect of diaphragmatic breathing exercise on urinary incontinence treatment. The secondary purpose was to compare the effect of pelvic floor muscle exercises and diaphragmatic breathing exercises on urinary incontinence women.

Design: Participants were randomized into two groups: pelvic floor muscle exercises (Group PFM n=20) and diaphragmatic breathing exercises (Group DB n=20). Exercise programs consisted of 1 set of contractions per day and each set included 30 repetitions for 6 weeks. Women were asked to complete forms of Incontinence Impact Questionnaire (IIQ-7) and the Urogenital Distress Inventory (UDI-6), Incontinence Quality of Life (I-QOL), and Overactive Bladder (OAB-V3) before starting the program and again at the end of the 6-week program. Changes from baseline were compared in both groups and between the two groups.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is a chronic condition with involuntary urine loss. Urgency urinary incontinence (UUI) is a complaint of involuntary loss of urine associated with urgency; stress urinary incontinence (SUI) is a complaint of involuntary urine leaks out on effort or physical exertion including sporting activities, or on sneezing or coughing. In the mixed type of urinary incontinence (MUI) complaints coexist both in stress and urgency.

Although urinary incontinence is not a life-threatening condition, the feeling of discomfort caused by constant wetness, irritation, and the fear of odor affects the daily and social activities of in patients.

The abdominal-pelvic cavity contains most of the internal organs, is bounded by the diaphragm above, abdominal muscles anterior and lateral, thoracolumbar fascia and dorsal muscles in the back, and pelvic floor in the lower part. The respiratory diaphragm forms the roof of the abdomina-pelvic cavity and the pelvic floor forms the base. The diaphragm is the main respiratory muscle, connected to the pelvic floor via the transversalis fascia. The pelvic floor supports internal organs, as well as constrictor and continence mechanisms of the urethral, anal and vaginal orifices in females.

Musculofascial support is provided by the pelvic floor forms a hammock onto which the urethra is compressed during increases in intra-abdominal pressure. When intraabdominal pressure increases, intra-abdominal contents downward momentum is arrested by stretch resistance of the pelvic floor structures. At this time, the proximal intraabdominal portion of the urethra is compressed against the underlying supporting layer, which consists of the endopelvic fascia, vagina, and pelvic floor.

Pelvic floor muscle (PFM) exercises, defined by Arnold H. Kegel, aims to regain support to the urinary organs by actively functioning the pelvic floor muscles. Previous researches show that PFM exercises are an effective treatment for UI and improve the quality of life (Qol) of in women. It is currently used as the first choice in conservative treatment of incontinence. However, PFM exercises may be encountered with some difficulties in order to understanding and performing by patients.

Talas et al. showed that the pelvic floor moves in the craniocaudal direction parallel to the diaphragm during respiration. In this study, they suggested that during expiration, the pelvic floor muscles contract together with the abdominal muscles, pushing the abdominal organs up, pushing the intra-abdominal pressure (IAP) to towards the diaphragm.

In this study, the investigators hypothesized that the patients can improve pelvic floor function by performing DB exercises, indirectly via the facial and functional connection between the diaphragm and PFM, and incontinence could be reduced.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of urinary incontinence
* Urinary leakage at least 3 months
* Not received physiotherapy before

Exclusion Criteria:

* Pregnancy
* Postpartum period (6 weeks after delivery)
* Detrusor hyperreflexia
* Menopause
* Hormonal therapy
* Active vaginal lesion or infection
* Urinary infection
* Prior pelvic surgery
* Organ prolapse
* Chronic pelvic pain
* Sexual disorders
* Neurological problem

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-16 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Incontinence Impact Questionnaire (IIQ-7) scores of women who performed diaphragmatic breathing exercises at 6 weeks | 6 weeks
  The Incontinence Impact Questionnaire (IIQ-7) is used to analyze the impact of UI on various activities and emotional states. Responses were on a 4-step ordered category scale from "not at all" to "greatly". Women were asked to complete those forms before starting the diaphragmatic breathing exercises and again at the end of the 6-week program.
Change from baseline the Urogenital Distress Inventory (UDI-6) scores of women who performed diaphragmatic breathing exercises at 6 weeks | 6 weeks
  The Urogenital Distress Inventory (UDI-6) is used to analyze the impact of UI on various activities and emotional states. Responses were on a 4-step ordered category scale from "not at all" to "greatly". Questions 1 and 2 of UDI-6 are directed to irritative symptoms, questions 3 and 4 address stress symptoms, others address obstructive or voiding symptoms. Women were asked to complete those forms before starting the diaphragmatic breathing exercises and again at the end of the 6-week program.
Change from baseline The Incontinence Quality of Life (I-QOL) scores of women who performed diaphragmatic breathing exercises at 6 weeks | 6 weeks
  The Incontinence Quality of Life (I-QOL) contains 22 items, on a 6 point Likert scale ranging from 0 (none) to 5 (very great deal), about limiting behaviors and social life impacts, low scores indicate poorer QoL. Women were asked to complete those forms before starting the diaphragmatic breathing exercises and again at the end of the 6-week program.
Change from baseline Overactive Bladder (OAB-V3) scores of women who performed diaphragmatic breathing exercises at 6 weeks | 6 weeks
  Overactive Bladder (OAB-V3) questionnaire consists of 8 questions about how bothered one is by symptoms of urinary urgency, urinary frequency, nocturia, ranging from never (0) to always (5). Women were asked to complete those forms before starting the diaphragmatic breathing exercises and again at the end of the 6-week program.

SECONDARY OUTCOMES:
Change from baseline Incontinence Impact Questionnaire (IIQ-7) scores of women who performed pelvic floor exercises at 6 weeks. | 6 weeks
  The Incontinence Impact Questionnaire (IIQ-7) is used to analyze the impact of UI on various activities and emotional states. Responses were on a 4-step ordered category scale from "not at all" to "greatly". Women were asked to complete those forms before starting the pelvic floor exercises and again at the end of the 6-week program.
Change from baseline Urogenital Distress Inventory (UDI-6) scores of women who performed pelvic floor exercises at 6 weeks. | 6 weeks
  The Urogenital Distress Inventory (UDI-6) is used to analyze the impact of UI on various activities and emotional states. Responses were on a 4-step ordered category scale from "not at all" to "greatly". Questions 1 and 2 of UDI-6 are directed to irritative symptoms, questions 3 and 4 address stress symptoms, others address obstructive or voiding symptoms. Women were asked to complete those forms before starting the pelvic floor exercises and again at the end of the 6-week program.
Change from baseline Incontinence Quality of Life (I-QOL) scores of women who performed pelvic floor exercises at 6 weeks. | 6 weeks
  The Incontinence Quality of Life (I-QOL) contains 22 items, on a 6 point Likert scale ranging from 0 (none) to 5 (very great deal), about limiting behaviors and social life impacts, low scores indicate poorer QoL. Women were asked to complete those forms before starting the pelvic floor exercises and again at the end of the 6-week program.
Change from baseline Overactive Bladder (OAB-V3) scores of women who performed pelvic floor exercises at 6 weeks. | 6 weeks
  Overactive Bladder (OAB-V3) questionnaire consists of 8 questions about how bothered one is by symptoms of urinary urgency, urinary frequency, nocturia, ranging from never (0) to always (5). Women were asked to complete those forms before starting the pelvic floor exercises and again at the end of the 6-week program.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol Universty, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hay-Smith EJC, Starzec-Proserpio M, Moller B, Aldabe D, Cacciari L, Pitangui ACR, Vesentini G, Woodley SJ, Dumoulin C, Frawley HC, Jorge CH, Morin M, Wallace SA, Weatherall M. Comparisons of approaches to pelvic floor muscle training for urinary incontinence in women. Cochrane Database Syst Rev. 2024 Dec 20;12(12):CD009508. doi: 10.1002/14651858.CD009508.pub2. PMID 39704322
- [Derived] Toprak N, Sen S, Varhan B. The role of diaphragmatic breathing exercise on urinary incontinence treatment: A pilot study. J Bodyw Mov Ther. 2022 Jan;29:146-153. doi: 10.1016/j.jbmt.2021.10.002. Epub 2021 Oct 20. PMID 35248263